CLINICAL TRIAL: NCT06865963
Title: Vestibulodynia At High Resolution: Omics Approach to Improve Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Barbara Gardella, Clinical professor, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 2022CLTAYH_002
Record Dates: First submitted 2025-03-01; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Vestibulodynia (VBD); Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — mRNA, protein, cells, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who receive diagnosis of vestibulodynia
  Interventions: Genetic: vulvar biopsy and blood semples
- patients without vulvar pain
  Interventions: Genetic: vulvar biopsy and blood semples

INTERVENTIONS:
Genetic: vulvar biopsy and blood semples — Collection of different types of specimen from VBD patients and healthy controls: mRNA, protein, cells, blood

SUMMARY:
According to recent nomenclature, vulvodynia is vulvar pain without a clear identifiable cause persisting for at least 3-months and distinguished from vulvar pain caused by a specific disorder (inflammatory, neoplastic, traumatic). Vulvodynia can be provoked (when the pain is felt after touching the area), or unprovoked (pain is constant). Localized provoked vulvodynia of the vestibule, known as vestibulodynia (VBD), is the most common manifestation of the disease (about 80%). Data collected suggests that up to 16% of women, particularly sexually active reproductive-aged women, suffers from this condition. Despite affecting almost 1 out of 8 women of all ages, vulvodynia remains completely unacknowledged to the most. These data highlight that VBD cannot be considered a rare disease, but it rather is a high frequency women's health condition, albeit neglected and hard to diagnose because of a lack of obvious markers. Despite the paucity of molecular data, studies about pathogenesis of VBD have highlighted several risk factors including inflammation, recurrent vulvovaginal infections and microbiota dysfunction, mucosal nerve fiber proliferation, hormonal alterations, pelvic floor muscle dysfunction, central pain mechanisms, and genetic factors. A recent study has highlighted that, compared to healthy controls, women with VBD demonstrated differences primarily in vaginal (but not plasma) concentrations of metabolites of the sphingolipid signaling pathways, suggesting localized effects in vagina and vulvar vestibule rather than systemic effects. The current prevalent theory on the etiology of VBD is that during or after an initial and persistent vulvovaginal insult (infection, microtrauma, allergic reaction), a "susceptible" individual is then unable to successfully clear the inflammation process that alters and sensitizes the neural tissue in the vestibular area, resulting in localized allodynia and hyperalgesia. The under-diagnosis of VBD is the result of different factors including practical, cultural, sociological and psychological ones. The women with VBD confirmed that healthcare provider knowledge and attitudes as well as system challenges (specialist and allied healthcare provider availability) are major barriers to timely diagnosis, mainly due to lack of diagnostic tests. For instance, many patients do not seek treatment due to feelings of inadequacy, invalidation, isolation or guilt. This attitude also has a cultural background that is rooted in shame, in the endurance of pain, in embarrassment and resulting silence of patients, dismissal of vulvar pain as a "psychological disorder" by clinicians have resulted in widespread ignorance about this disabling condition. Finally, one of the most important, and doubtlessly the easiest one to solve, is the lack of either molecular or cellular markers of the disease itself. Unfortunately the VBD diagnosis always comes too late, when the mechanism of aberrant immune response already has caused the irreversible nervous sprouting in the vulvar vestibule and the chronicization of the symptoms has already happened. This delayed diagnosis increases the women's risk for sexual dysfunction and diminishes their quality of life. The VBD diagnosis is generally a diagnosis of exclusion, where basically all other possible differential diagnoses have been excluded and this is what is "left over". Many markers of inflammation were investigated without significant results, likely because the method employed in the study was focused on few pre-selected targets and an unbiased analysis has not been performed, yet. For all these reasons, the search for suitable diagnostic markers of VBD remains a high but unmet research priority. In the NGS era the absence of genomic study of VBD is despicable. RNA-sequencing of vestibule vaginae (vestibular) cell swab is a pain-free method that we already tested and could allow the identification of diagnostic markers of VBD for the development and the optimization of a reliable and quantifiable diagnostic test. In this context we plan to perform transcriptomic analysis integrated with the state-of-the-art single cell omic analysis on VBD patients and healthy controls to unbiasedly identify specific VBD markers. Moreover, considering the different pathogenesis and the range of symptoms and severity of the disease, with these markers we also aim at stratifying different groups of VBD. This stratification will lay the foundation for further studies to move patients towards a real personalized medicine. This analysis has never been performed on VBD patients with this global approach and at such high resolution. The results of our project will help the clinicians in VBD diagnosis, in therapy direction and in the earlier identification of patients with higher risk to develop chronic VBD, thus helping to build a preventive strategy to avoid the progression and chronicization of the symptoms

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50
* abstinence from intercourse for 7 days prior to the visit
* non-use of intravaginal products for 7 days prior to the visit

Exclusion Criteria:

* patients whit generalized vulvodynia and those with only spontaneous, but not provoked vestibulodynia
* Endometriosis
* Pregnancy
* Infectious vulvar disease
* Post-menopause
* Feeding time
* gave birth within 4 months
* received systemic or vaginal antimicrobial or probiotic therapy within 1 month before the visit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who receive diagnosis of vestibulodynia.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Molecular marker: mRNA | 12 months
  identification of molecular markers, either at the mRNA expression, that can distinguish VBD patients from healthy controls and also distinguish different types of VBD patients

SECONDARY OUTCOMES:
Molecular marker: protein | 12 months
  identification of molecular markers, in particular proteins expression, that can distinguish VBD patients from healthy controls and also distinguish different types of VBD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Ostetricia e Ginecologia 1, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
at the end of the study
Supporting Information: Study Protocol